CLINICAL TRIAL: NCT04617964
Title: Intra and Interoperator Reproducibility of the Measurement of the Right Portal Vein Diameter at the Third Trimester Scan
Brief Title: Reproducibility of the Measurement of the Right Portal Vein Diameter
Acronym: PORTALGROWTH1
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020- A01910-39
Record Dates: First submitted 2020-10-13; First posted 2020-11-05 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Intrauterine Growth Retardation (IUGR)
Keywords: small-for-gestational-age; right portal vein; third-trimester ultrasound; intra and inter-operator reproducibility
MeSH Terms: conditions — Fetal Growth Retardation | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IUGR: sample of 40 pregnant women affected by intrauterine growth restriction (IUGR) Two referees will perform four successive measurements of the diameter of the right portal vein (RPV) during the same ultrasound examination at the third trimester. Each operator will qualify the appearance of the right portal vein as normal or collapsed using an evaluation grid, and will independently performe a series of two measurements using the same method.
  Interventions: Other: Ultrasound
- NORMAL: Ssample of 40 healthy pregnant women Two referees will perform four successive measurements of the diameter of the right portal vein (RPV) during the same ultrasound examination at the third trimester. Each operator will qualify the appearance of the right portal vein as normal or collapsed using an evaluation grid, and will independently performe a series of two measurements using the same method.
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Assessment the intra and interoperator reproducibility of the measurement of the right portal vein diameter at the routine third trimester ultrasound
  Other Names: Third trimester ultrasound

SUMMARY:
Although routine ultrasound is offered during the third trimester of pregnancy, less than a quarter of newborns with intrauterine growth retardation (IUGR) are suspected antenatally.

The measurement of the right portal vein (RPV) diameter on the transverse abdominal view at the 32 weeks' scan may be a new a tool for detecting small-for-gestational-age (SGA) at birth. The irregular and collapsed aspect of the right portal vein (RPV) on the third trimester ultrasound could be used for identifying hypoxemic and growth-restricted fetuses.

However, to our knowledge, the only interoperator reproducibility study of this measurement was performed using the same stored images or datasets without performing a new examination.

The main objective of this study is to assess the intra and interoperator reproducibility of the measurement of the right portal vein diameter at the routine third trimester ultrasound.

The secondary objective is to quantify the interoperator reproducibility of the assessment of the aspect, normal or collapsed, of the right portal vein, using an evaluation grid.

Two referees will perform four successive measurements of the diameter of the right portal vein (RPV) during the same ultrasound examination at the third trimester. Each operator will qualify the appearance of the right portal vein as normal or collapsed using an evaluation grid, and will independently performe a series of two measurements using the same method.

ELIGIBILITY:
Inclusion Criteria:

* Women carrying a pregnancy from 30 weeks to 33 weeks either normal or with IUGR,
* Patient without guardianship or curatorship or subordination,
* Patient benefiting from a Social Security scheme

Exclusion Criteria:

* Presence of a fetal malformation,
* Multiple pregnancy,
* Premature rupture of membranes,
* History of bariatric surgery,
* Body mass index (BMI)> 30 kg / m2,
* Patient benefiting from enhanced protection, namely: minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social establishment, adults under legal protection.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population comprise 80 consecutive pregnancies between 30 and 33 weeks, including 40 pregnant women with normal pregnancy, and 40 pregnant women affected by IUGR.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Measurement of the right portal vein diameter | Through study completion, an average of 1 year
  Intra and interoperator reproducibility of the measurement of the right portal vein diameter at the routine third trimester ultrasound

SECONDARY OUTCOMES:
Aspect of the right portal vein diameter | Through study completion, an average of 1 year
  Interoperator reproducibility of the assessment of the aspect, normal or collapsed, of the right portal vein, using an evaluation grid

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U. de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No